CLINICAL TRIAL: NCT00944697
Title: An Exploratory, Randomised, Double-blind, Single-dummy, Placebo Controlled, Parallel Group Study to Demonstrate the Analgesic Efficacy of Oxycodone/Naloxone Prolonged Release Tablets in Addition to Pregabalin Compared to Pregabalin Alone in Opioid-naïve Subjects Treated With Pregabalin Suffering From Moderate to Severe Pain Due to Diabetic Polyneuropathy
Brief Title: A Study to Demonstrate the Analgesic Efficacy of Oxycodone/Naloxone Prolonged Release Tablets in Addition to Pregabalin Compared to Pregabalin Alone in Opioid-naïve Subjects Treated With Pregabalin Suffering From Moderate to Severe Pain Due to Diabetic Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OXN2502; 2008-005815-17
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2012-02-28 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Moderate to Severe Pain Due to Diabetic Polyneuropathy
MeSH Terms: interventions — oxycodone naloxone combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablets (Placebo Comparator): A placebo tablet to match the active reference treatment
  Interventions: Drug: Placebo tablets
- Tablet (Active Comparator): Oxycodone Naloxone tablets
  Interventions: Drug: Oxycodone Naloxone

INTERVENTIONS:
Drug: Oxycodone Naloxone — Oxycodone Naloxone tablets
  Arms: Tablet
Drug: Placebo tablets — Placebo Oxycodone Naloxone tablets
  Arms: Tablets

SUMMARY:
To show superior analgesic efficacy of OXN PR in addition to a patient's current dose of pregabalin compared to pregabalin alone.

DETAILED DESCRIPTION:
Study OXN2502 is a pilot, exploratory, randomised, placebo-controlled, double-blind, single-dummy, parallel group study to assess efficacy and safety of OXN PR in addition to a patient's current dose of pregabalin compared to pregabalin alone in opioid-naïve subjects treated with pregabalin suffering from moderate to severe pain due to diabetic polyneuropathy.

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe pain due diabetic polyneuropathy
* Opioid-naive subjects

Exclusion criteria:

* Females who are pregnant or lactating
* Subjects with evidence of significant structural abnormalities of the gastrointestinal tract
* Subjects with evidence of impaired liver/kidney function upon entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Oliver Emrich, Ludwigshafen, Germany

REFERENCES:
- See also: Results available on website — http://www.mundipharma-rd.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was 13 July 2009 to 26 March 2010. There were 29 sites in General Practice, hospitals and SMOs.
Pre-assignment Details: Patients had to have moderate to severe pain due to diabetic/idiopathic polyneuropathy. This was shown by a pain score of >= 5 (average pain over 24 hours)and an MNSI (Michigan Neuropathy Screening Instrument) of >= 2.5 at screening. Subjects were then randomised to OXN (Oxycodone/Naloxone) or placebo.
Groups:
- Placebo Tablets: A placebo tablet to match the active reference treatment
- OXN PR Tablet: Oxycodone Naloxone Prolonged Release (OXN PR) tablets
Period: Overall Study
Arm/Group | Placebo Tablets | OXN PR Tablet
Started | 50 | 48
Completed | 48 | 43
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Administrative | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablets | OXN PR Tablet | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 35 | 67
  >=65 years | 18 | 13 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 62.24 (9.39) | 58.96 (10.03) | 60.63 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  Czech Republic | 21 | 19 | 40
  Germany | 7 | 7 | 14
  Hungary | 11 | 11 | 22
  Romania | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Short Form McGill Pain Score.
Description: The McGill Pain Score is the sum of the answers to three questions: A - describe your pain during the last week, 15 descriptors, (from 0 to 45 total), B - rate your pain during the last week (from 0 to 100), C: present pain intensity (0 to 5). Total pain score will be out of 150, with 0 being least pain and 150 being most pain.
Time Frame: Visit 2 (randomisation) and Visit 10 (end of study (12 weeks) or withdrawal)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Tablets | OXN PR Tablet
Number analyzed (Participants) | 50 | 46
units on a scale | 49.56 (29.62) | 47.65 (30.27)

ADVERSE EVENTS:
Time Frame: From after consent to 7 days after Last Patient Last Visit (105 days)
Description: Screening phase = 14 days, Treatment for 12 weeks (84 days) and 7 day follow up.
Arm/Group | Placebo Tablets | OXN PR Tablet
Serious Adverse Events (participants affected / at risk) | 0/50 | 4/48
Other Adverse Events (participants affected / at risk) | 22/50 | 36/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablets (N=50) | OXN PR Tablet (N=48)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) — This subject also had an SAE (Serious Adverse Event) of Iliac Artery Stenosis. Unrelated to study drug.
Iliac Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1) — This patient also had an SAE (Serious Adverse Event) of Coronary Artery Disease. Unrelated to study drug.
Cystitis (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to study drug.
Wound Abscess (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to study drug.
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — "Unlikely" relationship to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablets (N=50) | OXN PR Tablet (N=48)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 2
Ear and Labyrinth disorder (Ear and labyrinth disorders) | 4 | 3
Gastrointestinal Disorders (Gastrointestinal disorders) | 10 | 17
General Disorders and Administration Site Conditions (General disorders) | 1 | 7
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 (0) | 1
Infections and Infestations (Infections and infestations) | 3 | 9
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 | 0 (0)
Investigations (Investigations) | 6 | 6
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 4 | 3
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 0 (0)
Nervous System disorders (Nervous system disorders) | 5 | 12
Psychiatric Disorders (Psychiatric disorders) | 1 | 2
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 1
Respiratory, Thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 4
Vascular Disorders (Vascular disorders) | 0 (0) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No